CLINICAL TRIAL: NCT05771519
Title: Development and Assessment of an HIV Disclosure Intervention for Men in Uganda
Brief Title: Developing an HIV Disclosure Intervention for Men in Uganda
Acronym: DASH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Pooja R. Chitneni.,MD, Instructor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022P003409; K23MH126771 (NIH)
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: HIV Infections; Sexually Transmitted Infections (Not HIV or Hepatitis)
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Hepatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV disclosure intervention (Experimental): Participants assigned to the intervention group will likely participate in the following:
  * Sexual health education
  * Cognitive behavioral therapy strategies
  * Problem-solving skills building
  * Motivational interviewing
  * Developing a personalized HIV disclosure plan
  * Communication skills building
  * Role-playing disclosure strategies Procedures in both arms will encompass 3-5 individual sessions lasting 30-60 minutes over 2-3 months. There may also be a booster session at approximately the six-month timepoint.
  Interventions: Behavioral: HIV disclosure intervention
- Control (No Intervention): Participants assigned to the control group will likely participate in educational topics related to healthy living for men living with HIV. Procedures in both arms will encompass 3-5 individual sessions lasting 30-60 minutes over 2-3 months. There may also be a booster session at approximately the six-month timepoint.

INTERVENTIONS:
Behavioral: HIV disclosure intervention — This will be a biobehavioral intervention focused on helping men with HIV to disclose their HIV status to a personal confidant inclusive with specific focus on sexual partners.
  Arms: HIV disclosure intervention

SUMMARY:
The goal of this clinical trial is to test an HIV disclosure intervention that the investigators are developing focused on men living with HIV in Uganda. The main questions the investigators are trying to answer is whether the HIV disclosure intervention the investigators develop will help men who receive this intervention to disclose their HIV status to a greater extent than men who receive standard care.

Participants assigned to the intervention group will likely participate in the following:

* Sexual health education
* Cognitive behavioral therapy strategies
* Problem-solving skills building
* Motivational interviewing
* Developing a personalized HIV disclosure plan
* Communication skills building
* Role-playing disclosure strategies

ELIGIBILITY:
For all 3 Aims, "index participants" inclusion criteria will include:

* men living with HIV
* with sexually transmitted infection symptoms (e.g., urethral discharge, genital lesions)
* either not accessing antiretroviral therapy (per self-report109 and/or clinic documentation) or accessing antiretroviral therapy without HIV viral suppression
* age ≥18 years,
* with at least one sexual partner in the past three months

Aims 2 and 3 have the additional inclusion criteria:

* men living with HIV without HIV disclosure to at least one partner.

In Aims 2 and 3, male participants will be encouraged to invite sexual partners for enrollment. These "partner participants" will have the following inclusion criteria:

* age ≥18 years
* partnered with an enrolled man who reports HIV disclosure or plans for HIV disclosure with study support
* referred by the male participant.

Exclusion Criteria:

* an inability to speak the local language (Runyankole) or English
* an inability to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — All index participants will self-identify as male. Partner participants who men disclose to and bring into the study can be either male or female.
Enrollment: 70 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
HIV disclosure intervention acceptability | 6 months
  Of 35 intervention participants, ≥70% (25 participants) rate all 4 items on the Acceptability of Intervention Measure (a 5-point Likert scales) as "agree" or higher. I will also assess intervention acceptability through qualitative interviews with participants and counselors.
HIV disclosure intervention feasibility | 6 months
  Feasibility is defined by the Feasibility of Intervention Measure, intervention fidelity, and session completion. A) Feasibility of Intervention Measure: Of 35 intervention participants, ≥70% (25 participants) rate all 4 items on the Feasibility of Intervention Measure (a 5-point Likert scale) as "agree" or higher, B) Fidelity: Assuming a five-session intervention with 25% English-transcribed (44/175 sessions), intervention fidelity is attained when ≥70% (31 sessions) achieve ≥90% fidelity to the protocol adherence checklist, C) Session completion: Of the 35 intervention participants, ≥70% attend ≥50% of sessions. I will also assess intervention acceptability through qualitative interviews with participants and counselors.

SECONDARY OUTCOMES:
Index participant-reported disclosure | 6 months
  Index participant-reported disclosure (measured by an expanded disclosure measurement tool and a Center For AIDS Research-funded HIV Disclosure Processes Model Measurement Scale in development.
Partner participant HIV study site/clinic testing and counseling | 6 months
  The investigators will measure the percentage of partners that participants bring to clinic for HIV testing.
HIV viral suppression | 6 months
  Participant HIV viral suppression measured by nucleic acid amplification testing.

CONTACTS AND LOCATIONS:
Overall Officials: Pooja Chitneni, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

IPD SHARING:
Plan to Share IPD: No